CLINICAL TRIAL: NCT04714593
Title: A Clinical Study to Evaluate the Safety and Effectiveness of CD19- BCMA CAR - T Cells Immunotherapy in Patients With Relapsed or Refractory Acute B Lymphocytic Leukemia
Brief Title: Targeting CD19 and CD22 CAR-T Cells Immunotherapy in Patients With Relapsed or Refractory Acute B Lymphocytic Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanxi Province Cancer Hospital (Other)
Collaborators: Shanghai Ultra-T Immune Therapeutics Co. LTD (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T SXZL02
Record Dates: First submitted 2021-01-07; First posted 2021-01-19 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Acute Lymphocytic Leukemia， B-Cell
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: According to the sequence from the low dose group to the high dose group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose Group (Experimental): CD19-CD22 CAR-T cells injection, infused only once,3-6 subjects of low dose group will be intravenously infuse with 0.5×10^6 CAR+T cells/kg.
  Interventions: Biological: CD19-CD22 CAR-T cells
- Middle Dose Group (Experimental): CD19-CD22 CAR-T cells injection, infused only once,3-6 subjects of low dose group will be intravenously infuse with 2×10^6 CAR+T cells/kg.
  Interventions: Biological: CD19-CD22 CAR-T cells
- High Dose Group (Experimental): CD19-CD22 CAR-T cells injection, infused only once,3-6 subjects of low dose group will be intravenously infuse with 5×10^6 CAR+T cells/kg.
  Interventions: Biological: CD19-CD22 CAR-T cells
- Amplification Dose Group (Experimental): CD19-CD22 CAR-T cells injection, infused only once.After determined maximum tolerated dose,15 subjects of amplification dose group will be intravenously infuse with 0.5-5.0×10^6 CAR+Tcells/kg.
  Interventions: Biological: CD19-CD22 CAR-T cells

INTERVENTIONS:
Biological: CD19-CD22 CAR-T cells — A autologous doping CAR - T cells injection targets with CD19 and CD22，fluorine dara marina injection(30 mg/m2，QD×3d) and cyclophosphamide injection (300 mg/m2，QD×3d)will be used to remove the lymphocyte before infusion CD19-CD22 CAR-T cells .
  Other Names: Fluorine dara marina injection; Cyclophosphamide injection

SUMMARY:
Evaluation the safety,tolerability, preliminary efficacy,and PK/PD of CD19-CD22 CAR-T cells for the treatment of acute B lymphocytic leukemia.

DETAILED DESCRIPTION:
A non randomized study ,plans to enrollment 24 subjects of acute B lymphocytic leukemia .The subjects will divide into low, medium and high dose groups，to evaluate the safety and tolerability of CD19-CD22 CAR - T cells，to evaluate the preliminary efficacy and observe PK/PD parameters of CD19-CD22 CAR -T cells immunotherapy in patients with relapsed or refractory acute B lymphocytic leukemia .

ELIGIBILITY:
Inclusion Criteria:

1. 6-70 - year - old male or female subjects (including 6 years old and 70 years old, 6-18 subjects use only the recommended dose of treatment);
2. The Clinical diagnosis of recurrent/refractory acute B lymphocytic leukemia, after at least 2 courses of treatment, has not been achieved partial response, still in the continuous phase and progress, including the MRD positive, or recurrent intramedullary patients；
3. Bone marrow samples inspection by using flow cytometry or organization pathology ，the cell membrane surface antigen CD19 and/or CD22 positive；
4. ECOG physical status score of 0 to 2 points;
5. Expected lifetime is more than 12 weeks;
6. The clinical laboratory test results of screening phase meet the following criteria: (7 days before the inspection without blood transfusion) Hb≥60 g/L (allowed to use recombinant human erythropoietin); PLT≥ 50 x 10 ^ 9 / L ; ALC≥0.3×10^9/L; ANC≥0.75×10^9/L (allowed to use granulocyte colony stimulating factor); AST≤3ULN,ALT≤3ULN,TBIL≤2ULN；Ccr≥30 mL/min/1.73 m2；
7. Cardiopulmonary function: left ventricular ejection fraction > 40%; Baseline blood oxygen saturation > 95%;
8. Has a history of allogeneic/allogeneic hematopoietic stem cell transplantation patients: transplantation in 3 months ago, no grade 2 or more active graft versus host disease (GVHD), more than a month without immune inhibitors.

Exclusion Criteria:

1. The active hepatitis b, HBV - DNA detection lower limit of the subjects above research center; Hepatitis c virus (HCV) antibody positive and peripheral blood HCV - RNA positive subjects; Antibodies to HIV positive subjects; Early syphilis screening antibody positive;
2. The other clinical significance of active virus, bacterial infection, or failing to control systemic fungal infection;
3. Any instability of systemic disease, including but not limited to, unstable angina, cerebrovascular accident, or transient ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), New York heart association (NYHA) classification level III or higher congestive heart failure, drug control of serious arrhythmia, liver, kidney or metabolic diseases, as well as the standard treatment cannot control high blood pressure;
4. In past two years, because of autoimmune diseases such as crohn's disease, rheumatoid arthritis and systemic lupus erythematosus (sle), etc.) causing end-organ damage, or need systemic application of immunosuppressive drugs;
5. Had a history of the central nervous system diseases, such as epilepsy, serious brain damage, dementia, Parkinson's disease, psychosis,etc which influence the appraising of test,;
6. Diagnosed with other active malignancy in past five years(the basal or scaly skin cancer, superficial bladder cancer, breast cancer in situ, which has been cured and does not require follow-up treatment are not included );
7. Known allergic to cyclophosphamide, fluorine dara marina or CAR - T cell s including accessories, DMSO ;
8. Patients with pregnancy or lactation, patients do not want to take effective contraceptive measures within 6months after infusion CAR-T cells;
9. The other situations that researchers determined doesn't fit to participate in this study.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT | Form infusion CAR-T cells to 28 days after infusion
  Observe wether dose limiting toxicity will happened in dose escalation phase
ORR | Form infusion CAR-T cells to 2 years after infusion
  The overall response rate after CD19-CD22 CAR-T Cells immunotherapy

SECONDARY OUTCOMES:
Incidence of various types of adverse recation | Form infusion CAR-T cells to 2 years after infusion
  According to CTCAE 5.0, record the level , type of adverse events, evaluat the correlation of CD19-CD22 CAR-T cells
PFS | Form infusion CAR-T cells to 2 years after infusion
  Progression-free surial
DOR | Form infusion CAR-T cells to 2 years after infusion
  Duration of Response
OS | Form infusion CAR-T cells to subjects died，assessed up to 60 months
  Overall survival
Cmax | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  By measuring the CAR - T cells copy number and the positive rate, peak plasma concentration is determined
Tmax | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The maximum concentration of time
AUC（0-720d） | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  Area under the plasma concentration versus time curve
Concentration of IL2 level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（IL2 ）in peripheral blood
Concentration of IL6 level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（IL6 ）in peripheral blood
Concentration of IL10 level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（IL10 ）in peripheral blood
Concentration of TNF-α level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（TNF-α ）in peripheral blood
Concentration of IFN-γ level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（IFN-γ ）in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Liping Su, M.D., Principal Investigator — Hematology Department of ShanXi Cancer Hospital
Locations (1):
- Hematology Department of ShanXi Cancer Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Plan to Share Clinical Study Report within six months after the study completed
Supporting Information: CSR
Time Frame: Within six months after the study completed
Access Criteria: Research site